CLINICAL TRIAL: NCT04218253
Title: Clinical Application of Preoperative Nutritional Support Package for Liver Cancer
Brief Title: Clinical Application of Nutrition Support Package Before Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 20191226
Record Dates: First submitted 2019-12-29; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-10

CONDITIONS: Liver Neoplasms; Nutrition Therapy; Hepatectomy
Keywords: Nutrition Therapy; Hepatectomy
MeSH Terms: conditions — Liver Neoplasms | interventions — Amino Acids; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutritional intervention (Experimental): 300 or 500 calories nutritional support before operation according to the level of malnutrition
  Interventions: Dietary Supplement: 300 calories or 500 calories nutrient rich in branched chain amino acids and dietary fiber; Behavioral: Dietary mission
- control group (Other): Dietary education was conducted according to preoperative nutritional requirements
  Interventions: Behavioral: Dietary mission

INTERVENTIONS:
Dietary Supplement: 300 calories or 500 calories nutrient rich in branched chain amino acids and dietary fiber — 300 kcal rich in branched chain amino acids and water soluble dietary fiber (12g) for Mild malnutrition, or 500 kcal rich in branched chain amino acids and water soluble dietary fiber (12g) for moderate to severe malnutrition. The degree of malnutrition is determined by Patient-Generated Subjective Global Assessment (PG-SGA).
  Arms: nutritional intervention
Behavioral: Dietary mission — Dietary education was conducted according to preoperative nutritional requirements

SUMMARY:
Objective:To confirm the effect of preoperative oral nutrition therapy on patients with malnourished before liver cancer resection.

Study design:Prospective, randomized, controlled clinical study. Primary end point: incidence of all complications 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of primary liver cancer (including hepatocellular carcinoma, bile duct carcinoma, and mixed cell carcinoma)
* 2. No contraindications for surgery
* 3. Eastern Cooperative Oncology Group (ECOG) score of preoperative physical state <2 points
* 4. Preoperative liver function score Child-Pugh ≤ 6 points: total bilirubin ≤ 3.0 mg / dl, albumin ≥ 28 g / L, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤ 5 times the upper limit of normal
* 5. Voluntarily enter the study and sign the informed consent form, and communicate well with the researcher

Exclusion Criteria:

* 1. Patients who took fish oil supplements within 3 weeks before the study began
* 2. Patients with severe nutritional risk: serious nutritional risk should be considered when combining any of the following conditions: weight loss > 10% within 6 months; digital pain score (NRS) score > 5 points; BMI <18.5 kg/m2 (all patients with severe nutritional risk undergo individualized supportive care);
* 3. Patients with malignant tumors in other parts
* 4. Patients who are pregnant or lactating
* 5. Patients with mental and neurological disorders who cannot cooperate with medical staff
* 6. Patients with severe diabetes or poor glycemic control
* 7. Patients cannot tolerate nutritional preparations
* 8. Other circumstances that the researcher considers inappropriate to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications at 30 days after surgery | up to 30 days after surgery
  Postoperative complications were defined by Clavien-Dindo. Grade 1： Any deviation from the normal postoperative course without the need for pharmacologic treatment or surgical, endoscopic, and radiologic interventions. Allowed therapeutic regimens are drugs as antiemetics, antipyretics, analgetics, and diuretics, and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade 2： Requiring pharmacologic treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade 3： Requiring surgical, endoscopic, or radiologic intervention 3a： Intervention not under general anesthesia 3b： Intervention under general anesthesia Grade 4：Life-threatening complication (including CNS complications) requiring IC/ICU management.
  4a： Single organ dysfunction (including dialysis) 4b： Multiple organ dysfunction Grade 5： Death as a result of complications

SECONDARY OUTCOMES:
Postoperative hospital stay | up to 90 days after surgery
  from the date of the operation to the date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, Doctor, Study Chair — Tianjin Medical University cancer Instituteand Hospital
Locations (1):
- Tianjin Medical University cancer Instituteand Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided